CLINICAL TRIAL: NCT03292055
Title: Evaluation of the Psychometric Properties of a Food Frequency Questionnaire Developed for Patients With Coronary Heart Disease in Northern China
Brief Title: Food Frequency Questionnaire (FFQ) for Coronary Heart Disease (CHD) Patients
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Youjuan Zhang, Graduate Assistant, Chinese University of Hong Kong
Other Study IDs: 2016.557
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Coronary Heart Disease
Keywords: food frequency questionnaire; psychometric properties
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood testing for the blood glucose, lipid profile
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the psychometric properties of a newly developed FFQ specified for northern Chinese CHD and their high risk patients (CHD-FFQ). The psychometric properties include test-retest reliability, content validity, convergent validity, discriminant validity, concurrent validity and predictive validity. Particularly, this study will measure the physiological indicators, including plasma lipid profile (i.e. TG, TC, HDL-C, LDL-C), BG, BP and BMI twice at baseline and the end. The level of these physiological indicators will be compared with the fat intake measured by the CHD-FFQ, i.e. the baseline intake to test its convergent validity. It is also expected to predict the diet-related progression of CHD risks among high-risk individuals, i.e. patients with two or more CHD risk factors as following: raised fasting blood glucose (BG) level, increased blood pressure (BP), increased triglycerides (TG), decreased HDL-Cholesterol (HDL-C), increased LDL-Cholesterol (LDL-C), smoking and central obesity (International Diabetes Federation, 2015). In addition, this study will provide the FFQ's concurrent validity in assessing the intake of energy and nutrients against the CDC-FFQ. Moreover, whether the FFQ could detect the known differences in energy intake between men and women will be established for its discriminant validity.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* Have no CHD at enrollment;
* At high risk of CHD with at least two of the following risk factors:

  * current smoking: current smokers are defined as individuals who smoked regularly during the last 12 months
  * central obesity: for Chinese, central obesity is defined as waist circumstance above 90cm for male and 80cm for female, or with BMI above 30kg/m²
  * raised BP (systolic BP [SBP] ≥ 130 mmHg or diastolic BP [DBP] ≥85 mmHg or under antihypertensive treatment)
  * raised fasting BG (FBG) (100mg/dL [5.6mmol/L]) or under treatment with insulin or oral hypoglycemic agents
  * elevated TG (150mg/dL [1.7mmol/L])
  * elevated TC (≥ 240 mg/dL [5.18 mmol/L])
  * raised LDL-C (≥ 160 mg/dL [4.15 mmol/L])
  * decreased HDL-C (<40 mg/dL [1.03 mmol/L] for males, and <50 mg/dL [1.29 mmol/L] for females)
  * undergoing hyperlipidemia treatment

Exclusion Criteria:

* Impaired bilateral hearing
* Impaired mental status (according to their medical record)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CHD high-risk patients (corresponding to the inclusion criteria)
Sampling Method: Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Intake of Food | January-February, April- May, July- August, October- November
  The newly developed FFQ (CHD-FFQ) will be applied to the participants to collect their dietary intake of food.
Cardiac-related physiological blood parameters | January- February, October- November
  In the beginning and the end of the study, the medical records of the participants will be refered to get the blood glucose, total cholesterol, triglycerides, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol in the past three months, in the department and the community centers.
Height | January-February, April- May, July- August, October- November
  Participant's height will be measured to the nearest 0.5 cm, with a right-angle triangle resting on the scalp and against the wall, having the back square against the wall tape and eyes looking straight ahead. The height will be measured without wearing shoes.
Weight | January-February, April- May, July- August, October- November
  A calibrated scale with the resolution of 0.1 kg will be used to measure the weight of the participants, who will be asked to wear light clothes during measurement. The weight will be measured without shoes.
BMI | January-February, April- May, July- August, October- November
  weight and height will be combined to report BMI in kg/m^2
Waist circumstance | January-February, April- May, July- August, October- November
  Waist circumstance will be taken at the midpoint between the top of the iliac crest and the lower margin of the palpable rib
Blood pressure | January-February, April- May, July- August, October- November
  To take the blood pressure, the participant will be asked to be seated for at least 15 minutes with his/her legs uncrossed (WHO, 2008). Two BP measurements will be taken and between the two readings, the participant will have three minutes' rest.
Intake of Food | October-November
  As a criterion, the FFQ developed by Chinese CDC will be applied to the participants to collect their dietary intake of food.

SECONDARY OUTCOMES:
Sociodemographic information | January-February
  Age, gender, marital status, occupation, educational level, living conditions, financial background, and living areas will be collected using a self-developed questionnaire.
General clinical information | January-February
  Smoking history, family history and clinical data will be collected using a self-developed questionnaire.
Clinical Information | October- November
  Their clinical information on hospital readmission, surgery or medical procedures, and medication adjustment during the last year will be collected.
Physical activity level | January-February, April- May, July- August, October- November
  The physical activity level of the participants will be measured using the Chinese version of the short version of International Physical Activity Questionnaire (short- Chinese IPAQ).

CONTACTS AND LOCATIONS:
Overall Officials: SekYing CHAIR, PHD, Study Director — Chinese University of Hong Kong
Locations (2):
- China (2):
  - Qilu Hospital, Jinan, Shandong
  - Jinan Central Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No
All questionnaires and other collected data will be stored in a locked file cabinet, and no names or other personal data of participants will be used in publication. Only the PI and her supervisor will have access to these data.